CLINICAL TRIAL: NCT01474629
Title: Impact of Supplementation With Probiotics on Exercise-induced Oxidative Stress and Endotoxemia in Trained Men
Brief Title: Probiotic Sport Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Green Beat (Other)
Responsible Party: Principal Investigator, Lamprecht Manfred PhD, PhD, Principal investigator, Green Beat
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 23-509 ex 10/11
Record Dates: First submitted 2011-11-16; First posted 2011-11-18 (Estimated); Last update posted 2013-04-10 (Estimated); Status verified 2013-04

CONDITIONS: Oxidative Stress; Inflammation; Endotoxemia
Keywords: oxidative stress; inflammation; endotoxemia; strenuous exercise
MeSH Terms: conditions — Inflammation; Endotoxemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- probiotic-based dietary supplement (Active Comparator)
  Interventions: Dietary Supplement: probiotic-based dietary supplement
- placebo (Placebo Comparator)
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: probiotic-based dietary supplement — 24 trained men receive a probiotic-based dietary supplement for 16 weeks. Dosage 3x 10-9 per day
  Other Names: active group
  Arms: probiotic-based dietary supplement
Dietary Supplement: placebo — 24 trained men receive a placebo for 16 weeks with same dosage compared to active group
  Other Names: passive group
  Arms: placebo

SUMMARY:
We investigate the impact of a probiotic-based dietary supplement on oxidative stress and endotoxemia before and after strenuous exercise.

Hypotheses (H1):

* Supplementation has an influence on oxidative stress parameters before and post exercise
* Supplementation has an influence on parameters of endotoxemia and inflammation before and post exercise
* Strenuous exercise has an influence on parameters of oxidative stress, inflammation and endotoxemia

ELIGIBILITY:
Inclusion Criteria:

* trained men
* 30 - 45 years
* non-smokers
* 4wk wash out of all dietary supplements

Exclusion Criteria:

* untrained people (VO2max < 55 ml x kg-1)
* female
* all people not matching this age group
* smokers
* all men taking dietary supplements
* all men that fail in ergometric exercise eligibility testing, refering to the standards in sports medicine (e.g.: significant ST-decrease or increase, blood pressure > 240 mmHg, tachycardia, polymorphic extrasystolia, cyanosis, bradyarrhythmia..)
* all people that are not adjudged as "Healthy"

Ages: 30 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-10; Primary Completion 2012-03 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
markers of oxidative stress, endotoxemia and inflammation | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Lamprecht, PhD PhD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Graz, Austria

REFERENCES:
- [Derived] Lamprecht M, Bogner S, Schippinger G, Steinbauer K, Fankhauser F, Hallstroem S, Schuetz B, Greilberger JF. Probiotic supplementation affects markers of intestinal barrier, oxidation, and inflammation in trained men; a randomized, double-blinded, placebo-controlled trial. J Int Soc Sports Nutr. 2012 Sep 20;9(1):45. doi: 10.1186/1550-2783-9-45. PMID 22992437